CLINICAL TRIAL: NCT05862662
Title: Mobility Opportunities Via Education/Experience (MOVE): Healthcare Impact Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Center for Disability Services, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 21-003 Rev. B
Record Dates: First submitted 2023-04-13; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Quality of Life; Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children in MOVE Program: Children 5-12 years old who participated in the MOVE program for at least 12 continuous months prior to March 1, 2020 and again for at least 12 continuous months after August 2021.
  Interventions: Other: MOVE Program
- Adults in MOVE Program: Adults 22-65 years old who participated in the MOVE program for at least 12 continuous months prior to March 1, 2020 and again for at least 12 continuous months after August 2021.
  Interventions: Other: MOVE Program

INTERVENTIONS:
Other: MOVE Program — Mobility Opportunities Via Education functional therapy program.

SUMMARY:
The purpose of this study is to determine whether participation in the Mobility Opportunities Via Education (MOVE) program is associated with reduced use of healthcare for individuals with developmental disabilities.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether participation in the Mobility Opportunities Via Education (MOVE) program is associated with reduced use of healthcare for individuals with developmental disabilities. The investigators will compare healthcare "events" and healthcare expenditures for children and adults during intervals of at least one year when the subjects were participating in the MOVE program versus intervals of at least one year when the same individuals were not participating in the MOVE program based on health insurance records (i.e. Medicaid). Healthcare events are those which required professional medical services (associated with International Classification of Disease (ICD-XX) codes) or prescription medications. Healthcare events and healthcare expenditures will be reviewed from healthcare records obtained by Medicaid, Medicare, or private insurers and data will be compared between intervals.

ELIGIBILITY:
CHILDREN: Inclusion Criteria

* Males and females 5-21 years old.
* Participated in the MOVE program pre-COVID and post-COVID.
* Did not participate for at least 4 months in the MOVE program during COVID.
* Has a healthcare payor(s) who makes healthcare records available upon request.
* Subjects whose legal guardians are willing to give informed consent to obtain and review healthcare records from the subject's primary (and secondary, if applicable) payors.

CHILDREN: Exclusion Criteria

* Subjects who did not participate in the MOVE program through the duration of Interval #1 and Interval #3.
* Subjects whose legal guardians are unwilling to cooperate with the requests to obtain and review healthcare records and expenditures from the subject's primary (and secondary, if applicable) payors.

ADULTS: Inclusion Criteria

* Males and females 22-65 years old.
* Participated in the MOVE program during Interval #1 and Interval #3.
* Did not participate for at least 4 months in the MOVE program during Interval #2.
* Has a healthcare payor(s) who makes healthcare records available upon request.
* Subjects who are willing to give informed consent and/or subjects' legal guardians who are willing to give informed assent to obtain and review healthcare records from the subject's primary (and secondary, if applicable) payors.

ADULTS: Exclusion Criteria

* Subjects who did not participate in the MOVE program through the duration of Interval #1 and Interval #3.
* Subjects who are unwilling to give informed consent and/or subjects' legal guardians who are unwilling to give informed assent to cooperate with the requests to obtain and review healthcare records and expenditures from the subject's primary (and secondary, if applicable) payors.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with developmental disabilities who participated in the MOVE program for at least one year pre-COVID and are participating in the MOVE program post-COVID, but who did not participate in the MOVE program during COVID.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sum of Disability Adjusted Life Years | March 1, 2019 - April 30, 2023
  Healthcare events will be reviewed from the insurance record. International Classification of Disease (ICD) codes will be use to convert the healthcare event to disability adjusted life years. The sum of all disability adjusted life years will be calculated.
Number of Healthcare Events | March 1, 2019 - April 30, 2023
  Healthcare events will be reviewed from the insurance record. The number of visits for professional healthcare will be determined.
Cost of Healthcare Events | March 1, 2019 - April 30, 2023
  Healthcare events will be reviewed from the insurance record and total costs associated with healthcare utilization will be determined.
Cost of Medication Use | March 1, 2019 - April 30, 2023
  Insurance records will be reviewed and the cost of medication used will be determined.
Hip Range of Motion (Degrees) | March 1, 2019 - April 30, 2023
  From the Mobility Opportunities Via Education (MOVE) program records, hip range of motion (in degrees) will be determined.
PedsQL Quality of Life Scale Score | March 1, 2019 - April 30, 2023
  From the Mobility Opportunities Via Education (MOVE) program records, the Pediatric Quality of Life Inventory (PedsQL) outcome instrument will be used to determine quality of life. The PedsQL is comprised of 7 questions with each question scored on a scale of 0-4. Higher scores indicate a higher quality of life.
Top Down Motor Milestone Test Score | March 1, 2019 - April 30, 2023
  From the Mobility Opportunities Via Education (MOVE) program records, the Top Down Motor Milestone (TDMMT) score will be determined as an assessment of function

CONTACTS AND LOCATIONS:
Overall Officials: Eric H Ledet, Ph.D., Principal Investigator — Center for Disability Services
Locations (1):
- Center for Disability Services, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No